CLINICAL TRIAL: NCT05821088
Title: A Phase II Trial of Tafasitamab and Lenalidomide Followed by Tafasitamab and ICE as Salvage Therapy for Transplant Eligible Patients With Relapsed/ Refractory Large B-Cell Lymphoma
Brief Title: Tafasitamab and Lenalidomide Followed by Tafasitamab and ICE as Salvage Therapy for Transplant Eligible Patients With Relapsed/ Refractory Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Bond, MD (Other)
Responsible Party: Sponsor-Investigator, David Bond, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22140; NCI-2023-02612 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Recurrent B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classic Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Recurrent Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classic Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma, Not Otherwise Specified; Refractory Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Transformed Marginal Zone Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Specimen Handling; Carboplatin; Etoposide; Ifosfamide; Lenalidomide; Magnetic Resonance Spectroscopy; tafasitamab; Immunoglobulins; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tafasitamab, lenalidomide, ICE regimen) (Experimental): Patients receive tafasitamab IV, lenalidomide PO, etoposide IV, ifosfamide IV and carboplatin IV on study. Patients undergo PET or CT, and undergo blood sample collection throughout the study. Patients may undergo tissue biopsy on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Etoposide; Drug: Ifosfamide; Drug: Lenalidomide; Procedure: Positron Emission Tomography; Biological: Tafasitamab

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574

SUMMARY:
This phase II clinical trial evaluates tafasitamab and lenalidomide followed by tafasitamab and the carboplatin, etoposide and ifosfamide (ICE) regimen as salvage therapy for transplant eligible patients with large B-cell lymphoma that has come back (relapsed) or has not responded to treatment (refractory). Tafasitamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Lenalidomide may have antineoplastic activity which may help block the formation of growths that may become cancer. Drugs used in chemotherapy, such as carboplatin, etoposide and ifosfamide work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving tafasitamab and lenalidomide followed by ICE may be a better treatment for patients with relapsed or refractory large B-cell lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the anti-tumor activity of tafasitamab and lenalidomide followed by tafasitamab and ICE as first salvage therapy for relapsed/ refractory large B cell lymphoma as assessed by the cumulative complete response rate after completion of 2 or 4 cycles of study treatment.

SECONDARY OBJECTIVES:

I. Evaluate the overall response rate to tafasitamab and lenalidomide followed by tafasitamab and ICE in transplant eligible patients with relapsed/ refractory large B cell lymphoma after 2-4 total cycles of treatment.

II. Evaluate the overall and complete response rate to tafasitamab and lenalidomide after two cycles of treatment in transplant eligible patients with relapsed/ refractory large B cell lymphoma.

III. Evaluate the rate of successful stem cell mobilization following study treatment.

IV. Evaluate the rate of successful completion of autologous stem cell transplant (ASCT) following study treatment, including patients treated with a total of 2 or 4 cycles of treatment.

V. Evaluate the incidence of toxicities according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.

VI. Evaluate the progression free and overall survival in the study population. VII. Compare progression free survival (PFS)/ overall survival (OS) (i.e. long-term outcomes) in patients who proceed to transplant after completing only 2 cycles of tafasitamab/lenalidomide (tafa/len) versus those completing 4 cycles of tafa/len followed by tafa+ICE.

EXPLORATORY OBJECTIVES:

I. Evaluate the response rate to subsequent anti-CD19 CAR-T treatment in patients who go on to receive further therapy including for relapsed/ refractory disease.

II. Assess CD19 expression in patients with subsequent relapse or refractory disease following study treatment by immunohistochemistry.

III. Examine the association between clinical outcomes including complete response (CR) rate and pathological tumor characteristics (e.g. in activated B-cell [ABC]-type subgroup by gene expression profiling [GEP], non-germinal center [GC] subtype by Hans, "double/triple hit" phenotype by fluorescence in situ hybridization [FISH] and/or GEP).

IV. Examine the association between circulating tumor deoxyribonucleic acid (ctDNA) clearance and clinical outcomes including CR rate and PFS.

V. Evaluate association between clinical outcomes and duration of response to first-line therapy < 12 months vs > 12 months.

OUTLINE:

Patients receive tafasitamab intravenously (IV), lenalidomide orally (PO), etoposide IV, ifosfamide IV and carboplatin IV on study. Patients undergo positron emission tomography (PET) or computed tomography (CT), and undergo blood sample collection throughout the study. Patients may undergo tissue biopsy on study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 or older)
* Willing and able to provide written informed consent for the trial, assent when appropriate may be obtained per institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Considered transplant eligible by the treating physician
* Measurable disease by CT (defined as >= 1.5 cm in diameter) or one or more area of PET avid disease
* Have received one line of prior chemo-immunotherapy (i.e. cyclophosphamide, doxorubicin, prednisone, rituximab and vincristine [R-CHOP]). Note that corticosteroids for palliation of symptoms and radiation consolidation are not considered a line of therapy for purposes of eligibility determination
* Eligible histologic diagnosis includes: Diffuse large B cell lymphoma not otherwise specified (NOS), T cell histiocyte rich large B cell lymphoma, primary mediastinal B Cell lymphoma, follicular lymphoma grade 3B, high grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement, high grade B cell lymphoma NOS, DLBCL transformed from follicular lymphoma, DLBCL transformed from marginal zone lymphoma, DLBCL leg type, and B cell lymphoma unclassifiable (with features intermediate between DLBCL and classical Hodgkin's lymphoma)
* Absolute neutrophil count >= 1000 / mcL
* Platelets >= 75,000 / mcL in absence of transfusion support within 7 days of determining eligibility
* Hemoglobin >= 8.0 g/dL, with exception of cases in which cytopenias are due to marrow involvement by lymphoma
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL)
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 3.0 x ULN
* Serum creatinine clearance >= 60 mL/min (calculated according to institutional standard)
* Female subjects of childbearing potential should have a negative serum pregnancy test at screening and within 24 hours of receiving the first dose of study medication
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 3 months following the last dose of study treatment. Subjects should agree to ongoing pregnancy testing during the course of the study and after the end of study therapy. Subjects of childbearing potential are patients who have not been surgically sterilized and have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study therapy. Males must refrain from donating sperm during study participation and for 3 months after last dose of study medication
* In the opinion of the investigator, patients must be able and willing to receive adequate prophylaxis and/or therapy for thromboembolic events and be able to understand the reason for complying with the special conditions of the pregnancy prevention risk management plan
* Willing to provide archival tissue from biopsy performed after frontline systemic therapy (If prior archival tissue is unavailable, exceptions may be granted by the study principal investigator [PI])

Exclusion Criteria:

* Known active central nervous system involvement by lymphoma, including leptomeningeal involvement
* DLBCL transformed from chronic lymphocytic leukemia or small lymphocytic lymphoma (Richter's syndrome)
* Prior solid organ transplant
* Prior hematopoietic cell transplant
* History of other malignancy that could affect compliance with the protocol or interpretation of results in the opinion of the investigator
* Myocardial infarction or cerebrovascular accident within the past 6 months
* Clinically significant cardiovascular disease including uncontrolled arrhythmia or New York Heart Association Class 2-4 congestive heart failure
* Active uncontrolled infection or infection requiring IV antibiotic therapy
* Major surgery within 4 weeks prior to start of treatment other than surgery performed for diagnosis
* Prior lymphoma therapy should be completed greater than two weeks from the start of protocol therapy, with exception of patients receiving corticosteroids for palliation of symptoms
* Human immunodeficiency virus (HIV) infection AND CD4 count < 350 cells/ mm^3, evidence of resistant strain of HIV, or HIV viral load >= 50 copies HIV ribonucleic acid (RNA)/mL if on highly active antiretroviral therapy (HAART) or HIV viral load >= 10,000 copies HIV RNA/mL if not on anti-HIV therapy
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV DNA is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV RNA. Testing to be done only in patients suspected of having infections or exposures
* Known contraindication to any medication in the treatment plan, including known hypersensitivity
* Prior treatment with anti-CD19 targeted therapy or lenalidomide
* Gastrointestinal abnormalities including the inability to take oral medication, requirement of intravenous alimentation, or prior surgical procedure resulting in impaired enteral absorption of medication
* History or evidence of rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
* History of deep venous thromboembolism threatening thromboembolism, or known thrombophilia AND not willing to take venous thromboembolism prophylaxis during the study period
* Patients who in the opinion of the investigator have not recovered sufficiently from the adverse toxic events of prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | At the end of Cycle (each cycle is 28 days)
  Will be defined as patients who have achieved CR after two cycles (tafasitamab and lenalidomide) or four cycles as assessed by positron emission tomography (PET) imaging.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years
  Will be calculated with patients who achieve CR or partial remission (PR) at end of induction therapy as the numerator and all eligible patients who start treatment as the denominator, with a 95% binomial confidence interval provided.
Progression free survival | From start of treatment to progression or death, whichever occurs first, assessed up to 2 years
  Will be estimated by the method of Kaplan-Meier.
Incidence of adverse events | Up to 5 years
  Will be conducted through the review of toxicity data. All adverse events will be summarized by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 criteria, and tabulated across all patients who received any treatment with a focus on severe (grade 3+) adverse events and toxicities that are deemed at least possibly related to study treatment. The proportion of patients who go off treatment due to adverse events or those who refuse to continue treated for lesser toxicities will also be captured.
Tolerability of treatment | Up to 5 years
  Will be assessed through assessing the number of patients who required dose modifications and/or dose delays.

CONTACTS AND LOCATIONS:
Overall Officials: David A Bond, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu